CLINICAL TRIAL: NCT06563921
Title: PRObiotic Mixed With Exercise THErapy USe in MAFLD (PROMETHEUS in MAFLD)
Brief Title: RE and Probiotics in MAFLD/NAFLD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nicolaus Copernicus University (Other)
Collaborators: Medical University of Warsaw (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, DSc Paweł Zalewski, Prof., Nicolaus Copernicus University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAFLD_NAFLD_probiotics_RE
Record Dates: First submitted 2024-08-12; First posted 2024-08-21 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: NASH; NAFLD; MAFLD
Keywords: NASH; MAFLD; NAFLD; Probiotics; Resistance training; Gut microbiota; Hypertrophy training
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental: probiotics supplementation + physical exercise program (Experimental): Behavioral: physical exercise program in the form of a resistance/hypertrophy-oriented resistance program Dietary Supplement: probiotics supplementation
  Interventions: Behavioral: physical exercise programme; Dietary Supplement: probiotics supplementation
- Active Comparator: resistance/hypertrophy-oriented resistance program (Active Comparator): resistance/hypertrophy-oriented resistance program
  Interventions: Behavioral: physical exercise programme
- Placebo (Placebo Comparator): Supplementation with placebo
  Interventions: Dietary Supplement: placebo
- Active Comparator: probiotics supplementation (Active Comparator): Supplementation with probiotics
  Interventions: Dietary Supplement: probiotics supplementation

INTERVENTIONS:
Behavioral: physical exercise programme — resistance/hypertrophy-oriented resistance programme
  Arms: Active Comparator: resistance/hypertrophy-oriented resistance program; Experimental: probiotics supplementation + physical exercise program
Dietary Supplement: probiotics supplementation — probiotics supplementation
  Arms: Active Comparator: probiotics supplementation; Experimental: probiotics supplementation + physical exercise program
Dietary Supplement: placebo — placebo
  Arms: Placebo

SUMMARY:
This project aims to evaluate the roles of the autonomic nervous system (ANS) and gut microbiota as correlates of clinical improvement in metabolic dysfunction-associated fatty liver disease (MAFLD) and non-alcoholic fatty liver disease (NAFLD) in response to a therapeutic regimen comprising resistance exercise and probiotic supplementation. The primary objective is to investigate the effects of these non-pharmacological interventions on MAFLD/NAFLD and to identify patient phenotypes based on baseline ANS profiles and gut microbiota composition that predict clinical responses.

DETAILED DESCRIPTION:
The human microbiome, understood here as the collective community of microorganisms, their genetic material, and metabolic products that colonize the body from birth, is particularly concentrated in the gut. The gut microbiome, dominated primarily by anaerobic bacteria, encompasses thousands of species and millions of genes distributed among the major phyla: Firmicutes, Bacteroidetes, Actinobacteria, Proteobacteria, and Verrucomicrobia. Recent research has increasingly focused on the gut microbiome due to its dysbiosis being linked to numerous diseases that may be modifiable through diet, supplementation, or physical activity. Dysbiosis of the gut microbiome has also been implicated in MAFLD and NAFLD, which are the most prevalent liver diseases globally, affecting approximately 35% of the adult population, with this prevalence expected to rise. The gut-liver axis has been extensively studied in relation to MAFLD/NAFLD due to the bidirectional interactions between the gut microbiota and hepatic function. The portal vein, which supplies approximately 70% of the liver's blood flow, facilitates this interaction by connecting the intestines to the liver. Patients with NAFLD/MAFLD typically exhibit increased intestinal permeability compared to healthy individuals, thereby increasing the liver's exposure to gut-derived bacteria, endotoxins, bacterial products, and inflammatory mediators.

Probiotics, defined as live microorganisms that confer health benefits to the host, have been shown in previous studies to enhance the integrity of the intestinal barrier, regulate the gut microbiota, reduce intestinal permeability, and mitigate immune and metabolic disturbances. These effects are particularly relevant in patients with NAFLD/MAFLD, where probiotics have been observed to reduce hepatic steatosis and inflammation-related damage.

Physical exercise, particularly structured programs, has been demonstrated to significantly improve liver function in patients with NAFLD/MAFLD and positively modulate the gut microbiota. Exercise may attenuate the production of reactive oxygen species (ROS) and other oxidative agents in NAFLD by regulating antioxidant enzymes and anti-inflammatory mediators. Additionally, exercise interventions in these patients have been shown to improve blood lipid profiles, including triglycerides, cholesterol, AST, and ALT levels, offering substantial clinical benefits. Although the existing literature predominantly emphasizes aerobic training, this study seeks to compare the effects of resistance training and probiotic supplementation in patients with NAFLD/MAFLD and to assess potential changes in clinical outcomes. Furthermore, the study will explore the influence of baseline ANS and gut microbiota profiles on the patients' responses to these non-pharmacological therapies.

ELIGIBILITY:
Inclusion Criteria:

• NAFLD/MAFLD or NASH diagnosis

Exclusion Criteria:

* significant (structural) limitation of movement of the upper and/or lower limbs
* Not fluent in English or Polish
* Have participated in any trial or research project within 3 months
* history of following alternative diets within 3 months before the study or alternating diet during the trial,
* nervous system disorders
* cognitive function impairment and dementia
* pregnancy or nurturing
* significant (structural) limitation of movement of the upper and/or lower limbs
* osteoporosis/osteopenia
* unable to understand instructions
* receiving insulin
* unregulated diabetes
* stage 3 hypertension
* orthostatic intolerance
* chronic diseases of the cardiovascular system
* shift work
* those who will be found to have any concomitant liver disease
* Participants with liver steatosis and regular alcohol consumption of > 30 g/day
* anticoagulants/antiplatelet therapy, immunosuppressants, antibiotics, corticosteroids, valproic acid, amiodarone, tamoxifen.Medication use of steroids, methotrexate, metformin. Use of agents such as vitamin E, omega-3 fatty acids, or medications with evidence for effects on NAFLD (pioglitazone, GLP-1 analogs, dipeptidyl peptidase IV inhibitors, ursodeoxycholic acid)
* prolonged compromised immunity (e.g. recent cytotoxic chemotherapy, HIV infection with a CD4 count < 240)
* active or prior history of invasive malignancy (except for curatively treated in situ carcinomas [e.g., cervix] or non-melanoma skin cancer) unless a complete remission was achieved
* previous surgery (bariatric, gastric, intestinal resection)
* parenteral nutrition (TPN) for the last 6 months
* active thyroid disorder
* Cushing's syndrome
* anticoagulant therapy
* antibiotics in the 3 months before inclusion
* regular use of a probiotic or prebiotic supplement within 3 months before enrollment;
* inclusion in a drug interventional trial in the previous 3 months
* Known allergy to probiotics
* Any implanted battery operated device (i.e. AICD, pacemaker, loop recorder, cochlear implant)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2030-09-10 (Estimated); Study Completion 2036-09-10 (Estimated)

PRIMARY OUTCOMES:
Change in liver fat measured using MRI | 12 weeks
Changes in liver fibrosis (FIB-4 score) | 12 weeks

SECONDARY OUTCOMES:
changes in weight in kilograms using scale | 12 weeks
changes in body fat mass in kilograms measured using bioelectrical impedance method | 12 weeks
changes in free-fat mass in kilograms measured using bioelectrical impedance method | 12 weeks
changes in visceral fat level measured using bioelectrical impedance method | 12 weeks
HDL | 12 weeks
LDL | 12 weeks
AST | 12 weeks
ALT | 12 weeks

OTHER OUTCOMES:
autonomic nervous system function measured using Task Force Monitor | 12 weeks
changes in maximal strength measured in kilograms | 12 weeks
changes in RMR measured using CPET | 12 weeks
changes in the dynamics of glucose in response to standardized breakfast intake using continuous glucose monitoring | 12 weeks
changes in gut microbiota using fecal samples | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paweł Zalewski, Prof., Principal Investigator — Nicolaus Copernicus University, Poland; Lynette Hodges, PhD, Study Chair — Massey University, New Zealand; Beata Januszko-Giergielewicz, Assoc. Prof., Principal Investigator — Nicolaus Copernicus University, Poland; Maciej Słupski, Prof., Principal Investigator — Nicolaus Copernicus University, Poland; Karolina Skonieczna-Żydecka, Prof., Principal Investigator — Pomeranian Medical University in Szczecin, Poland; Agnieszka Cudnoch-Jędrzejewska, Prof., Study Chair — Warsaw Medical University, Poland; Sławomir Kujawski, PhD, Principal Investigator — Nicolaus Copernicus University, Poland; Joanna Słomko, Prof., Principal Investigator — Nicolaus Copernicus University, Poland; Monika Prylińska-Jaśkowiak, PhD, Principal Investigator — Nicolaus Copernicus University, Poland; Karl J. Morten, Prof., Principal Investigator — Oxford University, UK; Hanna Tabisz, MSc, Principal Investigator — Nicolaus Copernicus University, Poland; Beata Januszko-Giergielewicz, Prof., Principal Investigator — Nicolaus Copernicus University, Poland

IPD SHARING:
Plan to Share IPD: Undecided
Data would be shared upon a reasonable request from other researches. Requests could be made with a contact Authors after publication of papers on the collected data.